CLINICAL TRIAL: NCT01655576
Title: Effectiveness of Placental Drainage in the Third Stage of Labor: a Randomized Clinical Trial
Acronym: PLADRAINAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, MD pHD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLADRAINAGE; Pla1 (Registry Identifier: Placenta1)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2012-07

CONDITIONS: Management of Delivery
Keywords: drainage; pregnancy; active management; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine clamping (No Intervention): After delivery of the newborn, umbilical cord at mothers end, will be left clamped until delivery of the placenta.
- Placental drainage (Experimental): After delivery of the newborn, umbilical cord at mothers end, will be left unclamped until delivery of the placenta.
  Interventions: Procedure: Placental drainage

INTERVENTIONS:
Procedure: Placental drainage — After delivery of the newborn, umbilical cord at mothers end, will be left unclamped until delivery of the placenta.
  Arms: Placental drainage

SUMMARY:
The purpose of this study is to determine if placental drainage shortens third period of labor and reduces postpartum blood lost.

DETAILED DESCRIPTION:
The study aims to compare the effectiveness of placental drainage versus maintenance of maternal cord clamped end in the third stage of labor to reduce postpartum blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Low risk pregnant women
* Pregnancy at term
* Women at low risk for assisted labor / delivery and postpartum care.
* Live Fetus

Exclusion Criteria:

* Women under 18, mentally handicapped and indigenous;
* Women who agreed to participate signed the Informed Consent, but evolved to cesarean section or instrumental delivery by forceps;
* Instrumental Delivery by forceps or c-section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Duration of the third period of labor | Six hours
  Time from delivery of the baby to the delivery of the placenta

SECONDARY OUTCOMES:
Postpartum blood loss | 24 hours
  Volume of blood lost 24 hours after birth
PPH | 24 hours
  Postpartum hemorrhage
Need of uterotonics | 24 hours
  use of aditional uterotonics ( prophylkatic use not included)
Need of blood transfusions | until discharge
  Need of blood transfusions

CONTACTS AND LOCATIONS:
Locations (1):
- IMIP, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Vasconcelos FB, Katz L, Coutinho I, Lins VL, de Amorim MM. Placental cord drainage in the third stage of labor: Randomized clinical trial. PLoS One. 2018 May 2;13(5):e0195650. doi: 10.1371/journal.pone.0195650. eCollection 2018. PMID 29718920